CLINICAL TRIAL: NCT04530019
Title: Magnetic Resonance-Guided Brachytherapy Innovations in Gynecologic Cancer-Methods to Identify Remnant Tumor Versus Scar Tissue in Relation to Radiation Therapy
Brief Title: Brachytherapy Innovations in Gynecologic Cancer
Status: Withdrawn | Type: Observational
Why Stopped: The study never opened.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00244401
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MR Group: Following standard MRI-guided Brachytherapy, patients will have images analyzed for quantification of residual tumor versus fibrosis. We will pilot-test an endovaginal coil, a deflectable MR stylet, real-time planning software, and auto-segmentation of normal and tumor tissue.

SUMMARY:
In this pilot study, the investigators will test tools designed to more precisely identify, define and create a radiation treatment plan to tumor remnants as separate from fibrotic or normal tissue in a Magnetic Resonance (MR) simulator in the department of radiation oncology. The investigators will examine if this beneficial for tumor versus normal tissue delineation, will result in more precise tumor targeting with radiation in an efficient manner and whether there would be fewer toxicities.

DETAILED DESCRIPTION:
This study is a clinical research study following patients for toxicity after brachytherapy, and the investigators will be using the D2cc as a surrogate biomarker for determining risk for toxicity in addition to utilizing toxicity measured from physician-queries using the Common Toxicity Criteria for Adverse Events (CTCAE v. 4.0). Patients will have images analyzed for quantification of residual tumor versus fibrosis. The investigators will utilize Magnetic Resonance (MR) tracking, and pilot test: an endovaginal coil, a deflectable Magnetic Resonance stylet, real-time planning software, and auto-segmentation of normal tissues and tumor.

Standard T2-weighted MR images are generally recommended given the soft-tissue visualization without the need for contrast media injection. At the time of brachytherapy, acquisition of para-axial, para-sagittal and para-coronal images should be performed with the orientations being orthogonal (para-axial) and parallel (para-sagittal/para-coronal) to the intrauterine tandem. Slice thickness has a direct impact on applicator reconstruction accuracy, and a slice thickness of ≤3mm is required on the NRG Oncology study (NRG-GY006).

More advanced multi-parametric magnetic resonance imaging (mmpMRI) series show significant promise. A Dynamic Contrast Enhanced (DCE) study identified one voxel cluster consisting of low-enhancing voxels based on the relative signal increase (RSI) time series that was related to locoregional control (adjusted p-value 0.048). Diffusion-weighted (DW)-MRI is used to identify areas of dense residual tumor.31 In one analysis, the mean apparent diffusion coefficient (ADC) value of the primary tumor on pretreatment MRI was an independent predictor of disease-free survival in cervical cancer patients treated with chemoradiation. However, artifacts result in inconsistent contouring at the time of brachytherapy. 3D Slicer is a free open source software application for medical image computing, and will be utilized for some aspects of research in MR Simulator Suite.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

* Participants must have histologically or cytologically confirmed carcinoma. Central pathology review is not required; however, pathology will be reviewed at the Sidney Kimmel Comprehensive Cancer Center (SKCCC) at Johns Hopkins.
* Any patient eligible for internal implantation without MR guidance will be considered eligible for this protocol. Standard criteria for internal implantation include:

Carcinoma of the cervix: Stage I-IVA or vaginal recurrence Carcinoma of the uterus: Stage IIIB (vaginal involvement), inoperable, or vaginal recurrence Carcinoma of the vagina: Stage I-IVA or vaginal recurrence Carcinoma of the vulva: Stage I-IVA or recurrence Carcinoma of the urethra based on treating physician's discretion

* Patients who have received prior radiation or chemotherapy may be enrolled on this study.
* Age > 18 years. Children do not develop these malignancies and therefore are not considered candidates for this trial.
* Life expectancy of greater than 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance scale. ECOG status of <2, based on treating physician's discretion
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Absolute neutrophil count < 500 at the time of brachytherapy
* A history of metal in the head or eyes

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with gynecological cancer.
Study Population: Women with gynecological cancer, ages 18 and older.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity rates calculated for patients enrolled on this study | Up to 24 months post treatment
  Toxicity rates will be calculated using the Common Terminology Criteria for Adverse Events (CTCAE v. 4.0)

SECONDARY OUTCOMES:
Change in tumor as assessed by MRI | Prior to treatment/at diagnosis and post-brachytherapy treatment up to 14 days
  Compare changes in tumor based on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Akila Viswanathan, MD, Study Chair — Johns Hopkins, School of Medicine, Radiation Oncology